CLINICAL TRIAL: NCT05144360
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Atenas Association in the Treatment of Type II Diabetes Mellitus and Hypertension
Brief Title: Efficacy and Safety of Atenas Association in the Treatment of Type II Diabetes Mellitus and Hypertension
Acronym: ATENAS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategy review
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0220-ATENAS
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Hypertension Associated; Type II Diabetes Mellitus
Keywords: Hypertension; Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atenas association (Experimental): The study is triple-dummy. The patient must take 3 tablets once a day, as follows:
  1 tablet Atenas, oral;
  1 tablet empagliflozin placebo, oral;
  1 tablet telmisartan + amlodipine placebo, oral.
  Interventions: Drug: Atenas
- Empagliflozin + telmisartan + amlodipine (Active Comparator): The patient must take 3 tablets once a day, as follows:
  1 tablet Atenas placebo, oral;
  1 tablet empagliflozin, oral;
  1 tablet telmisartan + amlodipine, oral.
  Interventions: Drug: Atenas placebo

INTERVENTIONS:
Drug: Atenas — ATENAS 1 coated tablet, once a day EMPAGLIFLOZIN PLACEBO Empagliflozin placebo 1 coated tablet, once a day TELMISARTAN + AMLODIPINE PLACEBO Telmisartan + amlodipine 1 coated tablet, once a day
  Arms: Atenas association
Drug: Atenas placebo — Drug: EMPAGLIFLOZIN Empagliflozin 25 mg 1 coated tablet, once a day. Drug: TELMISARTAN Telmisartan + Amlodipine 40 + 5/80 +5 mg 1 coated tablet, once a day ATENAS PLACEBO Atenas placebo 1 coated tablet, once a day
  Arms: Empagliflozin + telmisartan + amlodipine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Atenas association in the treatment of type 2 diabetes mellitus and hypertension

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants of both sexes, with age greater than or equal to 18 years and less than or equal to 85 years;
* Participants presenting the diagnosis of type II diabetes mellitus, and who did not reach the therapeutic goals of HbA1c with previous dietary, physical exercise guidance and previous therapies at a stable dose in the last 3 months;
* Participants presenting the diagnosis of hypertension, and who did not reach the therapeutic goals with previous therapies.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Known hypersensitivity to any of the formula compounds;
* Type 1 diabetes mellitus;
* Known or suspected secondary hypertension.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 120 days
  Changes from baseline in glycated hemoglobin
Systolic blood pressure (SBP) | 120 days
  Changes from baseline in SBP in ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Adverse events | 150 days
  Incidence and severity of adverse events recorded during the study